CLINICAL TRIAL: NCT04019613
Title: Assessment of Pulmonary Congestion During Cardiac Hemodynamic Stress Testing
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was stopped due to funding and time constraints.
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Brandon M. Wiley, M.D., Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 19-002499
Record Dates: First submitted 2019-06-28; First posted 2019-07-15 (Actual); Results first posted 2022-07-20 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-06

CONDITIONS: Dyspnea; Heart Failure With Preserved Ejection Fraction
Keywords: dyspnea; heart failure with preserved ejection fraction; pulmonary edema; lung ultrasound; extravascular lung water
MeSH Terms: conditions — Dyspnea; Pulmonary Edema

STUDY DESIGN:
Intervention Model Description: All patients undergoing a clinically indicated invasive cardiac hemodynamic exercise test will be eligible for enrollment into the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Subjects undergoing clinical invasive hemodynamic stress test (Experimental): Subjects scheduled for standard-of-care, clinically indicated, invasive hemodynamic stress test will undergo lung ultrasound and assessment of extravascular lung water by pulmonary thermodilution technique.
  Interventions: Diagnostic Test: Lung ultrasound

INTERVENTIONS:
Diagnostic Test: Lung ultrasound — Lung ultrasound will be performed at baseline (resting), prior to exercise with passive leg elevation, after 1.5 minutes of 20 Watts exercise, during each subsequent stage, at peak workload and at 1 minute recovery. Pulmonary thermodilution will be performed at rest, peak stress and at 1 minute recovery.
  Other Names: Pulmonary Thermodilution

SUMMARY:
The aim of this study is to utilize lung ultrasound to detect the development of extravascular lung water in patients undergoing clinically indicated invasive hemodynamic exercise stress testing for symptomatic shortness of breath. The study will correlate the lung ultrasound findings with cardiac hemodynamics and measurements of extravascular lung water in an effort to better understand the pathophysiology of exertional dyspnea.

DETAILED DESCRIPTION:
Exercise induced elevation of left ventricular (LV) filling pressures can be the source of chronic dyspnea. Ultimately, high LV filling pressure leads to the development of extravascular lung water (EVLW) which can cause symptoms of dyspnea. Lung ultrasound (LUS) is a highly feasible, non-invasive procedure that is extremely sensitive for detecting EVLW. The sonographic signature of EVLW is a reverberation artifact called a "B-Line". The study will evaluate the etiology of sonographic B-Lines using invasive hemodynamic catheterization while simultaneously measuring the amount of EVLW present during exercise stress testing using transpulmonary thermodilution. The study aim is to demonstrate that the severity of EVLW, assessed by number of B-Lines, will correlate with LV filling pressures. In addition, the study will test the hypothesis that patients demonstrating dynamic increases in sonographic B-Lines with exercise will also display more severe symptoms of dyspnea, altered ventilatory mechanics (higher ratio of minute ventilation to carbon dioxide production (VE/VCO2)), and reduced aerobic capacity (lower peak oxygen consumption (VO2)).

ELIGIBILITY:
Inclusion Criteria:

* All adult patients (≥18 years) who are referred for invasive cardiac hemodynamic assessment
* Patients who have the capacity to understand and consent for the research study

Exclusion Criteria:

* Patients with known interstitial lung disease or pulmonary fibrosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2019-11-08 (Actual); Primary Completion 2019-12-19 (Actual); Study Completion 2019-12-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barry Borlaug, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Subjects Undergoing Clinical Invasive Hemodynamic Stress Test
Started | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Subjects Undergoing Clinical Invasive Hemodynamic Stress Test
Number analyzed (Participants) | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.75 (17.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Correlation of the Number of Lung Ultrasound B-Lines With Intra-cardiac Filling Pressures
Description: Lung ultrasound will be performed during invasive stress testing. The number of B-lines visible during stress testing will be correlated with synchronous measurements of intra-cardiac filling pressures .
Time Frame: Lung ultrasound imaging for B-Lines and assessment of intracardiac hemodynamics will be performed during the scheduled invasive stress test (initial visit, day #1).
Population: Study terminated due to funding and time constraints. Data not collected or analyzed.
Arm/Group | Subjects Undergoing Clinical Invasive Hemodynamic Stress Test
Number analyzed (Participants) | 0

2. Secondary Outcome: Correlation of the Number of Lung Ultrasound B-Lines With Ventilatory Mechanics.
Description: Lung ultrasound will be performed during invasive stress testing. The number of B-lines visible during stress testing will be correlated with synchronous measurements ventilatory mechanic parameters measured using expiratory gas.
Time Frame: Lung ultrasound imaging and assessment of ventilatory mechanics (using analysis of expired gas) will be performed during the scheduled invasive stress test (initial visit, day #1).
Population: Study terminated due to funding and time constraints. Data not collected or analyzed.
Arm/Group | Subjects Undergoing Clinical Invasive Hemodynamic Stress Test
Number analyzed (Participants) | 0

3. Secondary Outcome: Correlation of the Number of Lung Ultrasound B-Lines Developed During Invasive Stress Testing With Measurement of Extravascular Lung Water.
Description: Lung ultrasound will be performed during invasive stress testing. The number of B-lines visible during stress testing will be correlated with synchronous measurements extravascular lung water using transpulmonary thermodilution.
Time Frame: Lung ultrasound imaging and assessment of the amount of extravascular lung water using transpulmonary thermodilution will be performed during the scheduled invasive stress test (initial visit, day #1).
Population: Study terminated due to funding and time constraints. Data not collected or analyzed.
Arm/Group | Subjects Undergoing Clinical Invasive Hemodynamic Stress Test
Number analyzed (Participants) | 0

4. Secondary Outcome: Lung Ultrasound B-Lines Developed During Invasive Stress and the Calculated Amount of Extravascular Lung Water Will be Correlated With Changes in the Levels of Serum Protein, Hemoglobin and Brain Natriuretic Peptide Levels.
Description: Lung ultrasound will be performed during invasive stress testing. The number of B-lines visible during stress testing will be correlated with synchronous measurements extravascular lung water using transpulmonary thermodilution. In addition, serum levels of hemoglobin, protein and brain natriuretic peptide will be collected, synchronously, during the stress test.
Time Frame: Serum biomarkers, lung ultrasound and assessment of extravascular lung water will be performed during the scheduled invasive stress test (initial visit, day #1).
Population: Study terminated due to funding and time constraints. Data not collected or analyzed.
Arm/Group | Subjects Undergoing Clinical Invasive Hemodynamic Stress Test
Number analyzed (Participants) | 0

5. Secondary Outcome: Correlation of the Number of Lung Ultrasound B-Lines Developed During Invasive Stress Testing With Clinical Outcomes.
Description: Lung ultrasound will be performed during invasive stress testing. The number of B-lines visible during stress testing will be correlated with patient clinical outcomes defined as a composite outcome of hospital readmission, non-fatal myocardial infarction, or cardiovascular death.
Time Frame: 24 months post-stress test.
Population: Study terminated due to funding and time constraints. Data not collected or analyzed.
Arm/Group | Subjects Undergoing Clinical Invasive Hemodynamic Stress Test
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from baseline to end of study participation for a total of approximately 1 day on all participants.
Arm/Group | Subjects Undergoing Clinical Invasive Hemodynamic Stress Test
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-28): https://cdn.clinicaltrials.gov/large-docs/13/NCT04019613/Prot_SAP_000.pdf